CLINICAL TRIAL: NCT03433131
Title: An Open Label Expanded Access Program Intended to Provide Treatment With HBS-101 (Pitolisant) to Adult Patients in the U.S. With Excessive Daytime Sleepiness Associated With Narcolepsy With or Without Cataplexy
Brief Title: Expanded Access Program to Provide Treatment With Pitolisant to Adult Patients in the U.S. With Excessive Daytime Sleepiness Associated With Narcolepsy With or Without Cataplexy
Status: No longer available | Type: Expanded Access
Sponsor: Harmony Biosciences Management, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HBS-101-CL-001
Record Dates: First submitted 2018-02-07; First posted 2018-02-14 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Narcolepsy Without Cataplexy; Narcolepsy With Cataplexy
MeSH Terms: conditions — Narcolepsy | interventions — pitolisant

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Pitolisant — Tablets
  Other Names: Wakix

SUMMARY:
This EAP will be open to provide access to treatment with pitolisant while a U.S. New Drug Application (NDA) is being prepared and submitted for review for marketing approval. This program will be open to adult patients in the U.S. with Excessive Daytime Sleepiness (EDS) associated with narcolepsy, with or without cataplexy. Pitolisant will be made available through treating physicians participating in the program.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the treating physician, the patient is capable of understanding and complying with protocol and program requirements, oral drug administration and care instructions.
2. The patient or, when applicable, the patient's legally acceptable representative, signs and dates a written, ICF and any required privacy authorization prior to the initiation of any program procedures.
3. Men or women, 18 years of age and over.
4. Patients with a diagnosis of narcolepsy with or without cataplexy according to the ICSD or DSM criteria at the time of diagnosis.
5. Patients should be free of prohibited treatments or have discontinued them for at least 7 days prior to the start of treatments.
6. Women of child-bearing potential must have a negative serum pregnancy test performed at the screening visit.
7. Due to the effectiveness of hormonal contraceptives potentially being reduced when used with pitolisant, alternative or concomitant barrier methods of contraception are required for patients taking hormonal contraceptives (e.g., ethinyl estradiol) when taking pitolisant and for at least 21 days after discontinuation of pitolisant treatment.

Exclusion Criteria:

1. The patient has severe hepatic impairment (Child-Pugh C).
2. The patient is a woman who is breastfeeding or plans to breastfeed during their participation.
3. The patient has, in the judgment of the treating physician, a history or current medical condition that could affect safety or poses an additional risk to the patient by their participation in the program.
4. The patient is at high risk for suicide defined as a suicide attempt within the past year, significant risk determined by the investigator interview, or use of the Columbia Suicide Severity Rating Scale (C-SSRS).
5. The patient has a history of hypersensitivity or allergic reaction to pitolisant or any inactive ingredient of the formulation.
6. Current or recent (within one year) history of a substance abuse or dependence disorder including alcohol abuse as defined in Diagnostic and Statistical Manual of Mental Disorders (DSM-V).
7. Patients with a known history of long QTc syndrome (e.g. syncope or arrhythmia) or any significant history of a serious abnormality of the ECG (e.g. recent myocardial infarction), or QTc Fridericia higher than 450 ms for male and 470 ms for female (electrocardiogram Fridericia's corrected QT interval = QT / 3√ RR).
8. Significant abnormality in the physical examination or clinical laboratory results.
9. Prior severe adverse reactions to CNS stimulants.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Michael Thorpy, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (69):
- United States (69):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - CPC, Cullman, Alabama
  - Xenoscience, Phoenix, Arizona
  - Foothills Neurology, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Sleep Medicine Specialists of California, San Ramon, California
  - Santa Monica Sleep Disorders Center, Santa Monica, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Colorado Sleep Institute, Boulder, Colorado
  - Norwalk Hospital Sleep Disorders Center, Norwalk, Connecticut
  - Clinical Neurosciences fo Tampa Bay, Clearwater, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Sleep Medicine Specialists of South Florida, PA, Miami, Florida
  - Child Lung, Asthma Sleep Specialists, Winter Park, Florida
  - Emory University, Atlanta, Georgia
  - NeuroTrials Research Center, Atlanta, Georgia
  - The Neurological Center of North Georgia, Gainesville, Georgia
  - Critical Healthcare Decisions, Savannah, Georgia
  - Northwestern Medical Group, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - NorthShore Uni HealthSys-Glenbrook Hospital, Glenview, Illinois
  - Northshore Sleep Medicine, Northbrook, Illinois
  - Indiana Internal Medicine Consultants, Greenwood, Indiana
  - The University of Kansas Health System, Fairway, Kansas
  - Norton Pulmonary Specialists, Louisville, Kentucky
  - Maine Medical Partners - Neurology, Scarborough, Maine
  - The Center for Sleep and Wake Disorders, Chevy Chase, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - The University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Novi, Michigan
  - Bronson Sleep Health, Portage, Michigan
  - Alliance Health Shelby Family Medicine, Shelby, Michigan
  - Fairview Health Services, Brooklyn Park, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - St. Lukes Hospital, Sleep Medicine, Chesterfield, Missouri
  - University of Missouri, Columbia, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Norwell Health, New Hyde Park, New York
  - NYU-FGP Comphrenhensive Epilepsy Center-Sleep Center, New York, New York
  - Columbia University, New York, New York
  - Unity Sleep Disorders Center, Rochester, New York
  - University of Rochester Sleep Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Excel Psychiatric Associates, PA, Huntersville, North Carolina
  - Raleigh Neurology Assoc., PA, Raleigh, North Carolina
  - Neurology & Neuroscience Associates, Inc., Akron, Ohio
  - Intrepid Research, LLC, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Legacy Medical Group Sleep Medicine, Portland, Oregon
  - Collegeville Family Practice, Berwyn, Pennsylvania
  - Paoli Sleep Center, Paoli, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Maria J. Sunseri, MD, LLC, Pittsburgh, Pennsylvania
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Respitory Specialists, Wyomissing, Pennsylvania
  - Brown Medicine/Rhode Island Hospital, West Warwick, Rhode Island
  - Bogan Sleep Consultants, Columbia, South Carolina
  - Sleep Medicine Associates of Texas, Dallas, Texas
  - Houston Neurology & Sleep Center, Houston, Texas
  - Sleep Therapy & Research Center, San Antonio, Texas
  - Comprehensive Sleep Medicine Associates, Sugar Land, Texas
  - Chalottesville Neurology and Sleep Medicine, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Stultz Sleep and Behavioral Health, Barboursville, West Virginia
  - Medical College of Wisonsin, Milwaukee, Wisconsin

REFERENCES:
- See also: Program website to provide information to both prosective patients and physicians — http://thepeacenarcolepsyprogram.com